CLINICAL TRIAL: NCT01592604
Title: An Optimal Treatment for Avulsion Fractures of the Base of Fith Metatarsal Bone. A Level I Prospective Randomised Control Trial
Brief Title: An Optimal Treatment for Avulsion Fractures of the Base of Fith Metatarsal Bone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STH 15761
Record Dates: First submitted 2012-04-05; First posted 2012-05-07 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Closed Fracture of Base of Fifth Metatarsal Bone
Keywords: fracture; fifth metatarsal; functioanl outcome
MeSH Terms: conditions — Fractures, Bone

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment A (Experimental): Patients receive supportive compressive bandage for 4 weeks
  Interventions: Device: Compressive bandage
- Treatment B (Experimental): Below knee walking plaster cast for 4 weeks
  Interventions: Device: Below knee walking cast

INTERVENTIONS:
Device: Compressive bandage — Compressive below knee bandage for 4 weeks in group A
  Arms: Treatment A
Device: Below knee walking cast — Below knee walking cast for 4 weeks
  Arms: Treatment B

SUMMARY:
Avulsion fractures of the base (tuberosity) of fifth metatarsal bone are the most common fractures in the foot, frequently treated in fracture clinics and involving significant resources. At present methods of treatment and follow up vary widely from no active treatment to surgery, depending entirely on a treating doctor preference. There is no agreement on simple, safe and reliable method of treatment. The investigators believe that vast majority of these injuries heal well on its own without any specific treatment. By comparing two most commonly used treatments the investigators aim to establish one simple, safe and reliable mode of treatments. The investigators are going to evaluate functional results of these two treatments in a short and longer time prospective, by using the best available scientific tools. The investigators believe that results of the investigators study will eventually lead to change of practise and more efficient NHS care for these patients. It will reduce unnecessary treatments and clinic appointments, and bring substantial savings to the NHS in a long prospective.

DETAILED DESCRIPTION:
This is a randomised prospective control trial. Patients with these fractures will normally first come to the Emergency Department (ED), where they have a foot radiograph confirming a fracture, and initial treatment only. This treatment is arbitrary, depends on the assessing clinician preference and usually varies from supportive tight bandage or a supportive plaster cast with crutches. All of these patients are normally referred to an orthopaedic fracture clinic. It is an orthopaedic trauma clinician in the fracture clinic who determines and takes the responsibility for the definitive management of patients with this injuries and may decide to change the treatment initiated by the ED staff.

The investigators will inform clinical staff in the ED of the trial.The investigators will provide ED clinicians with patient information sheets. Patients who have this information sheet provided by the ED will have between a few hours and more than 24 hours "cool off" period to consider the information depending on next fracture clinic availability. Then they will be recruited in the fracture clinic should they wish to participate. The investigators must stress, however, that due to the nature of the ED service - high staff turn around, time pressure and other reasons beyond our control it is not possible to guarantee that all patients with relevant injuries will receive an information sheet in ED and have this "cool off" period to consider participation in. In such situations patients will be offered the information sheet, counselled and recruited, if they wish to, on their first presentation to the fracture clinic. The investigators believe that due to practical issues related to ED service this will be the likely situation for a significant proportion of patients. The investigators think this is an unavoidable situation.

Patients will be recruited on their first presentation to a fracture clinic should they consent. Using centralised electronic remote randomisation method patients will be allocated either to group A(symptomatic treatment)- double tubigrip and crutches with recommendation to weight bear as comfortable in normal footwear, or group B (active treatment) - below knee walking plaster cast with crutches and recommendation to weight bear as comfortable. This means that for many patients the initial treatment they received in ED will be changed but this often happens in normal current practice. Two treatment modes used in our study - supportive bandage and walking cast are the ones most commonly used normally. Patients declining to participate in the study will be treated and followed up according to patient and treating clinician preference and this also reflects the current practice. This study therefore deviates little from the current common practice. Patients in group B will be evaluated for venous thrombo-embolism (VTE) risk according to Sheffield Teaching Hospitals NHS Foundation Trust policy. Those whose risk is high will be offered anti-thrombotic prophylaxis according to the Trust policy for the duration of cast immobilization (4 weeks). Those patients will be counselled on benefits and risks of anti-thrombotic prophylaxis. On the whole we do not anticipate many patients to require anti-thrombotic prophylaxis.

Outcome measures: Primary outcome - foot functional outcome. We will use a Visual -Analogue-Scale Foot and Ankle (VAS FA) score. This is the only validated functional foot and ankle score. Secondary outcome - A) Health status and functional outcome, - Euroqol (EQ- 5D) - a standardised instrument for use as a measure of a health outcome and B) - foot function - American Foot and Ankle Society Foot and Ankle functional (AOFAS) score. This foot and ankle score is not validated, but most frequently used in the research literature. Additional outcomes will be records of unexpected return with the same problem, change of treatment modality, re-injury of the same foot and complications of treatment. The investigators will evaluate outcomes at four time points. Firstly, patients will complete baseline VAS FA, AOFAS, and EQ-5D questinnaires providing the level of functional impairment/disability prior to treatment. Patients in both groups will be seen in clinic at 4 weeks - at this stage cast will be removed in group B. At this point VAS FA, AOFAS, and EQ-5D questionnaires will be filled by patients in both groups in clinic. To see whether method of treatment has an effect in longer prospective the investigators will evaluate outcomes at 3 and 6 months. We anticipate that by this time fractures will heal uneventfully in the vast majority of patients . We believe that majority of patients is unlikely to return to clinic after such a long time. For this reason the investigators will post questionnaires to patients in both groups to be filled at home and posted back to us in confidential prepaid envelopes one week before their respective 3 and 6 month follow up. If a patient will decide to withdraw, or we have no response, - no further attempts to contact will be made. The investigators believe that this will save unnecessary follow up appointments, and also yield more results. In case of any problems all patients will be able to return to a fracture clinic for a help. The investigators will ask all patients in both groups to stop using crutches whenever they feel like to.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (older than 15 years of age) with an acute closed isolated type I avulsion fractures of the base of the fifth metatarsal bone, (within 7 days of the injury)

Exclusion Criteria:

* Diabetes, Inflammatory arthritis, previous same foot tarso-metatarsal fractures, previous same foot surgery, more than 7 days since the injury.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Validated Visual analague scale for foot and ankle (VAS FA) score | 6 months post treatment
  To evaluate functional outcome 6 months post treatment

SECONDARY OUTCOMES:
Euroqol 5D | baseline, 4 weeks, 3 months, 6 months post treatment
  Standardised general health functional outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Pavel - Akimau, MBChB, Principal Investigator — Sheffield Teaching Hopsitals
Locations (1):
- Northern General Hospital, Sheffield, South Yorkshire, United Kingdom